CLINICAL TRIAL: NCT01672983
Title: A Phase 2 Study to Evaluate the Safety, Tolerability, Antiviral Activity, and Pharmacokinetics of ABT-450 With Ritonavir (ABT-450/r) and ABT-267 in Japanese Adults With Chronic Hepatitis C Virus Infection
Brief Title: A Study to Evaluate ABT-450 With Ritonavir (ABT-450/r) and ABT-267 in Japanese Adults With Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M12-536
Record Dates: First submitted 2012-07-27; First posted 2012-08-27 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2015-10

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Japanese; Hepatitis C; Genotype 2; Genotype 1b; paritaprevir; ombitasvir; ritonavir; VIEKIRAX Combination Tablets
MeSH Terms: conditions — Hepatitis C | interventions — ombitasvir; paritaprevir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm 1 (Experimental): Participants with HCV GT1b received ABT-450/ritonavir (100/100 mg) and ABT-267 (25 mg) once daily for 12 weeks.
  Interventions: Drug: ABT-450/ritonavir, ABT-267
- Arm 2 (Experimental): Participants with HCV GT1b received ABT-450/ritonavir (150/100 mg) and ABT-267 (25 mg) once daily for 12 weeks.
  Interventions: Drug: ABT-450/ritonavir, ABT-267
- Arm 3 (Experimental): Participants with HCV GT1b received ABT-450/ritonavir (100/100 mg) and ABT-267 (25 mg) once daily for 24 weeks.
  Interventions: Drug: ABT-450/ritonavir, ABT-267
- Arm 4 (Experimental): Participants with HCV GT1b received ABT-450/ritonavir (150/100 mg) and ABT-267 (25 mg) once daily for 24 weeks.
  Interventions: Drug: ABT-450/ritonavir, ABT-267
- Arm 5 (Experimental): Participants with HCV GT2 received ABT-450/ritonavir (100/100 mg) and ABT-267 (25 mg) once daily for 12 weeks.
  Interventions: Drug: ABT-450/ritonavir, ABT-267
- Arm 6 (Experimental): Participants with HCV GT2 received ABT-450/ritonavir (150/100 mg) and ABT-267 (25 mg) once daily for 12 weeks.
  Interventions: Drug: ABT-450/ritonavir, ABT-267

INTERVENTIONS:
Drug: ABT-450/ritonavir, ABT-267 — ABT-450 (tablet) dosed with ritonavir (capsule), and ABT-267 (tablet)
  Other Names: ABT-450 also known as paritaprevir; ABT-267 also known as ombitasvir; ritonavir also known as Norvir; ABT/450/r/ABT-267 (ABT-450 coformulated with ritonavir and ABT-267) also known as VIEKIRAX Combination Tablets

SUMMARY:
This study evaluated the safety, tolerability, antiviral activity, and pharmacokinetics of ABT-450 (also known as paritaprevir) with ritonavir (ABT-450/r) and ABT-267 (also known as ombitasvir) in adult Japanese patients with chronic hepatitis C virus genotype 1b (HCV GT1b) or genotype 2 (HCV GT2) infection who were previous treated with pegylated interferon/ribavirin (pegIFN/RBV).

DETAILED DESCRIPTION:
This multicenter, randomized, open-label, parallel-arm, combination treatment study consisted of a Treatment and Post-treatment Phase, divided into 2 cohorts: 1) chronic HCV GT1b- infected, pegIFN/RBV treatment-exposed Japanese adults; and 2) HCV GT2-infected, pegIFN/RBV treatment-exposed Japanese adults. The Treatment Phase evaluated the antiviral activity, safety, and pharmacokinetics of a range of ABT-450/r and ABT-267 doses for 12 to 24 weeks. The Post-treatment Phase evaluated the evolution and persistence of viral resistance to ABT-267 and ABT-450.

ELIGIBILITY:
Inclusion Criteria:

* Females must be practicing specific forms of birth control on study treatment, or be post-menopausal for more than 2 years or surgically sterile
* Chronic hepatitis C, genotype 1b (HCV-GT1b) or genotype 2 (HCV GT2) infection (HCV RNA level greater than 10,000 IU/mL at screening) previously treated with pegylated interferon/ribavirin (pegIFN/RBV).
* Subject's hepatitis C virus genotype is subgenotype 1b and subject was a null responder or partial responder, OR
* Subject's hepatitis C virus genotype is subgenotype 2 and subject was a null responder, partial responder, or relapser (Null responder: received at least 10 weeks of pegIFN/RBV for the treatment of HCV and failed to achieve a 2 log10 IU/mL reduction in HCV RNA at Week 12; Partial responders: received at least 20 weeks of pegIFN/RBV for the treatment of HCV and achieved ≥ 2 log10 IU/mL reduction in HCV RNA at Week 12, but failed to achieve HCV RNA undetectable (HCV RNA < lower limit of detection [< LLOD]) at the end of treatment; Relapsers: received at least 1 course of pegIFN/RBV for the treatment of HCV and was undetectable at the end of treatment, but HCV RNA was detectable within 24 weeks of treatment follow-up).

Exclusion Criteria:

* Significant liver disease with any cause other than HCV as the primary cause
* Positive screen for drugs or alcohol.
* Positive hepatitis B surface antigen or anti-human immunodeficiency virus antibody.
* Use of contraindicated medications within 2 weeks of dosing
* Previous use of any investigational or commercially available anti-Hepatitis C virus agent other than pegIFN/RBV, including previous exposure to ABT-450 or ABT-267.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takuma Matsuda, MS, Study Director — AbbVie

REFERENCES:
- [Result] Chayama K, Notsumata K, Kurosaki M, Sato K, Rodrigues L Jr, Setze C, Badri P, Pilot-Matias T, Vilchez RA, Kumada H. Randomized trial of interferon- and ribavirin-free ombitasvir/paritaprevir/ritonavir in treatment-experienced hepatitis C virus-infected patients. Hepatology. 2015 May;61(5):1523-32. doi: 10.1002/hep.27705. Epub 2015 Mar 23. PMID 25644279
- [Derived] Schnell G, Tripathi R, Krishnan P, Beyer J, Reisch T, Irvin M, Dekhtyar T, Setze C, Rodrigues L Jr, Alves K, Burroughs M, Redman R, Chayama K, Kumada H, Collins C, Pilot-Matias T. Resistance characterization of hepatitis C virus genotype 2 from Japanese patients treated with ombitasvir and paritaprevir/ritonavir. J Med Virol. 2018 Jan;90(1):109-119. doi: 10.1002/jmv.24923. Epub 2017 Sep 22. PMID 28842997
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Started | 18 | 18 | 19 | 18 | 19 | 18
Completed Study Drug | 18 | 17 | 18 | 18 | 12 | 17
Completed | 18 | 18 | 19 | 18 | 19 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were summarized by treatment arm for all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6 | Total
Number analyzed (Participants) | 18 | 18 | 19 | 18 | 19 | 18 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (15.06) | 54.8 (11.96) | 61.9 (8.14) | 57.5 (10.15) | 62.5 (8.34) | 62.8 (7.89) | 59.2 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 12 | 10 | 12 | 10 | 59
  Male | 10 | 11 | 7 | 8 | 7 | 8 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks After Treatment (SVR24)
Description: The percentage of participants with SVR24 (plasma Hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantitation [< LLOQ] 24 weeks after the last dose of study drug). The LLOQ for the assay was 25 IU/mL.
Time Frame: 24 weeks after last dose of study drug
Population: Intent-to-treat (ITT) population: all subjects who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Number analyzed (Participants) | 18 | 18 | 19 | 18 | 19 | 18
percentage of participants | 100 [81.47 to 100.00] | 88.9 [65.29 to 98.62] | 100 [82.35 to 100.00] | 100 [81.47 to 100.00] | 57.9 [33.50 to 79.75] | 72.2 [46.52 to 90.31]

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence, which does not necessarily have a causal relationship with treatment. A serious adverse event (SAE) is an AE that results in death, is life-threatening, results in or prolongs hospitalization, results in congenital anomaly, persistent or significant disability/incapacity, spontaneous or elective abortion, or requires intervention to prevent a serious outcome. AEs were rated for severity as either Mild: transient and easily tolerated; Moderate: causes discomfort and interrupts usual activities; or Severe: causes considerable interference with usual activities, may be incapacitating or life-threatening. AEs related to study drug were assessed as being either probably or possibly related by the investigator. Treatment-emergent AEs (TEAEs) were collected from the first dose of study drug administration to 30 days after last dose; SAEs were collected from the time that informed consent was obtained to 30 days after last dose.
Time Frame: TEAEs: up to 16 weeks for the 12-week treatment groups and up to 28 weeks for the 24-week treatment groups; SAEs: up to 65 weeks for the 12-week treatment groups and up to 77 weeks for the 24-week treatment groups.
Population: Safety population: all participants who received at least 1 dose of study drug
Measure: Number; unit: participants
Groups:
- Arm 1 + Arm 5: Arm 1: Participants with HCV GT1b received ABT-450/ritonavir (100/100 mg) and ABT-267 (25 mg) once daily for 12 weeks; Arm 5: Participants with HCV GT2 received ABT-450/ritonavir (100/100 mg) and ABT-267 (25 mg) once daily for 12 weeks.
- Arm 2 + Arm 6: Arm 2: Participants with HCV GT1b received ABT-450/ritonavir (150/100 mg) and ABT-267 (25 mg) once daily for 12 weeks; Arm 6: Participants with HCV GT2 received ABT-450/ritonavir (150/100 mg) and ABT-267 (25 mg) once daily for 12 weeks.
Arm/Group | Arm 1 + Arm 5 | Arm 2 + Arm 6 | Arm 3 | Arm 4
Number analyzed (Participants) | 37 | 36 | 19 | 18
participants
  Adverse Events | 28 | 31 | 16 | 15
  Serious Adverse Events | 1 | 2 | 2 | 0

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Treatment (SVR12)
Description: The percentage of participants with SVR12 (plasma HCV RNA level < LLOQ 12 weeks after the last dose of study drug). The LLOQ for the assay was 25 IU/mL.
Time Frame: 12 weeks after last dose of study drug
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm 1: Hepatitis C Virus (HCV), genotype 1b (GT1b) participants received 100/100 mg ABT-450/ribavirin and 25 mg ABT-267 daily for 12 weeks.
- Arm 2: Hepatitis C Virus (HCV), genotype 1b (GT1b) participants received 150/100 mg ABT-450/ribavirin and 25 mg ABT-267 daily for 12 weeks.
- Arm 3: Hepatitis C Virus (HCV), genotype 1b (GT1b) participants received 100/100 mg ABT-450/ribavirin and 25 mg ABT-267 daily for 24 weeks.
- Arm 4: Hepatitis C Virus (HCV), genotype 1b (GT1b) participants received 150/100 mg ABT-450/ribavirin and 25 mg ABT-267 daily for 24 weeks.
- Arm 5: Hepatitis C Virus (HCV), genotype 2 (GT2) participants received 100/100 mg ABT-450/ribavirin and 25 mg ABT-267 daily for 12 weeks.
- Arm 6: Hepatitis C Virus (HCV), genotype 2 (GT2) participants received 150/100 mg ABT-450/ribavirin and 25 mg ABT-267 daily for 12 weeks.
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Number analyzed (Participants) | 18 | 18 | 19 | 18 | 19 | 18
percentage of participants | 100 [81.47 to 100.00] | 88.9 [65.29 to 98.62] | 100 [82.35 to 100.00] | 100 [81.47 to 100.00] | 57.9 [33.50 to 79.75] | 72.2 [46.52 to 90.31]

4. Secondary Outcome: Percentage of Participants With End of Treatment (EOT) Response
Description: The percentage of participants with EOT response (plasma HCV RNA level < LLOQ at week 12 for the 12-week duration arms and Week 24 for the 24-week duration arms12). The LLOQ for the assay was 25 IU/mL.
Time Frame: 12 or 24 weeks after first dose of study drug
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Number analyzed (Participants) | 18 | 18 | 19 | 18 | 19 | 18
percentage of participants | 100 [81.47 to 100.00] | 100 [81.47 to 100.00] | 100 [82.35 to 100.00] | 100 [81.47 to 100.00] | 63.2 [38.36 to 83.71] | 83.3 [58.58 to 96.42]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs (TEAEs) were collected from first dose of study drug administration to 30 days after last dose (up to 28 weeks); SAEs were collected from the time that informed consent was obtained to 30 days after last dose (total up to 77 weeks).
Description: TEAEs were collected from the first dose of study drug to 30 days after last dose (12-week treatment: up to 16 weeks; 24-week treatment: up to 28 weeks); SAEs were collected from the time that informed consent was obtained to 30 days after last dose (12-week treatment: total up to 65 weeks; 24-week treatment: total up to 77 weeks).
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Serious Adverse Events (participants affected / at risk) | 0/18 | 2/18 | 2/19 | 0/18 | 1/19 | 0/18
Other Adverse Events (participants affected / at risk) | 14/18 | 15/18 | 16/19 | 15/18 | 14/19 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=18) | Arm 2 (N=18) | Arm 3 (N=19) | Arm 4 (N=18) | Arm 5 (N=19) | Arm 6 (N=18)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
FLUID RETENTION (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=18) | Arm 2 (N=18) | Arm 3 (N=19) | Arm 4 (N=18) | Arm 5 (N=19) | Arm 6 (N=18)
HYPOCHROMIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
NEUTROPHILIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
PALPITATIONS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
ASTHENOPIA (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
BLEPHARITIS (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
CHALAZION (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0
DIPLOPIA (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
DRY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
PUNCTATE KERATITIS (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
STRABISMUS (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
DENTAL CARIES (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 0 | 0
DUODENAL ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 2
ENTERITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
ENTEROCOLITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
GINGIVAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
GLOSSODYNIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 2 | 0
RADICULAR CYST (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
CHEST DISCOMFORT (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
FATIGUE (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
MALAISE (General disorders) | 2 | 0 | 1 | 1 | 1 | 0
OEDEMA (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 0 | 0 | 2 | 1
PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
PYREXIA (General disorders) | 1 | 0 | 2 | 0 | 1 | 0
BILIARY COLIC (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0
SEASONAL ALLERGY (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 1
BRONCHITIS (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1
CYSTITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 2 | 2 | 2 | 0
GASTROENTERITIS BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
GINGIVITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
HELICOBACTER GASTRITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 1 | 6 | 4 | 9 | 5 | 7
PERIODONTITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
ARTHROPOD STING (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 0 | 1 | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
BLOOD BILIRUBIN UNCONJUGATED INCREASED (Investigations) | 1 | 0 | 1 | 1 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
BLOOD PRESSURE INCREASED (Investigations) | 1 | 0 | 0 | 1 | 0 | 1
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
PROTEIN URINE PRESENT (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
URINE LEUKOCYTE ESTERASE POSITIVE (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 2 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
MYOFASCIAL PAIN SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
AUTONOMIC NERVOUS SYSTEM IMBALANCE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
CERVICAL RADICULOPATHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
HEAD DISCOMFORT (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 2 | 1 | 3 | 1 | 3 | 5
MIGRAINE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
SOMNOLENCE (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
DYSPHORIA (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
INSOMNIA (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
NOCTURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
PROTEINURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
OROPHARYNGEAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
ALOPECIA AREATA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
CUTANEOUS LUPUS ERYTHEMATOSUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 1 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3 | 0 | 1
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
HOT FLUSH (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 1 | 2 | 2 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.